CLINICAL TRIAL: NCT03946566
Title: The Establishment and Analysis of the Clinical Prediction Model of Acupuncture and Moxibustion for Stroke Recovery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Yang Huiting, physician, The Third Affiliated hospital of Zhejiang Chinese Medical University
Other Study IDs: MRJ-HT-1001
Record Dates: First submitted 2019-05-07; First posted 2019-05-10 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Acupuncture Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acupuncture group: Using acupuncture, electric acupuncture, moxibustion and acupoint injection treatment.
  Interventions: Procedure: Acupuncture
- Basic treatment group: Use basic treatments, such as western medicine.
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Using acupuncture, electric acupuncture, moxibustion and acupoint injection treatment.

SUMMARY:
Electronic health records of stroke convalescent patients will be selected from the third affiliated hospital of Zhejiang Chinese Medical University from January 2012 to December 2019. Relevant clinical data will be extracted according to case data, and model-based decision tree analysis will be conducted to establish and evaluate the clinical prediction Model.

DETAILED DESCRIPTION:
Cases will be screened according to inclusion and exclusion criteria.Patients' basic information, risk factors, types of stroke, TCM diagnosis, all treatment during hospitalization, neurological impairment evaluation, imaging examination results and other contents will be recorded.Finally, statistical processing will be carried out to establish the prediction model, draw ROC curve and evaluate the model.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stroke
* The incidence is between 30 days and 180 days
* Age ≥ 18 years old
* The first onset

Exclusion Criteria:

* Subarachnoid hemorrhage
* transient ischemic attack
* other intracranial lesions
* Non-atherosclerotic thrombotic cerebral infarction
* Surgery, trauma, congenital disability leading to limb dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be stroke convalescent patients from The Third Affiliated Hospital of Zhejiang Chinese Medical University from January 2012 to December 2019.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Neurological Functional Impairment Assessment for Stroke Patients | Change from neurological functional impairment score at 6 months(or the last discharge time ，which less than 6 months)
  To evaluate the consciousness, muscle power, dysarthria, sensory disturbancen and ataxia of stroke patients on the first day, the seventh day, the fifteenth day, the first month and the sixth month after admission (or the last time of discharge).The total score is 0-29 points. The lower the score, the less the neurological defect. The efficacy will be assessed as an improvement in the neurological functional impairment score (eg, score improvement = score at admission - score at discharge), and treatment was effective when the score was reduced by more than 18%.

CONTACTS AND LOCATIONS:
Overall Officials: Ruijie Ma, Doctor, Study Director — The Third Affiliated hospital of Zhejiang Chinese Medical University
Locations (1):
- The Third Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China